CLINICAL TRIAL: NCT01096251
Title: Systemic and STRATegic Psychotherapy for OBesity
Brief Title: STRATOB: a Randomized Controlled Clinical Trial of Cognitive Behavioural Therapy and Brief Strategic Therapy With Telecare for Binge-eating Disorder
Acronym: STRATOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Gianluca Castelnuovo, prof., Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCAU-STRATOB-1
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Binge Eating Disorder
Keywords: Obesity; Binge Eating Disorder; Cognitive Behavioural Therapy; Brief Strategic Therapy; Telepsychology
MeSH Terms: conditions — Obesity; Binge-Eating Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Experimental): CBT group: in-hospital treatment (diet, physical activity, dietitian counseling, 8 sessions of CBT) plus 8 outpatient telephone-based sessions of CBT-oriented psychological support and monitoring with the same CBT inpatient psychotherapists.
  Interventions: Behavioral: CBT vs BST
- BST (Experimental): BST group: in-hospital treatment (diet, physical activity, dietitian counseling, 8 sessions of BST) plus 8 outpatient telephone-based sessions of BST-oriented psychological support and monitoring with the same BST inpatient psychotherapists.
  Interventions: Behavioral: CBT vs BST

INTERVENTIONS:
Behavioral: CBT vs BST — The comparison between the CBT and BST will be assessed in a two-arm randomized controlled trial. Participants will be randomly allocated in 2 groups (CBT and BST).

SUMMARY:
The STRATOB study is a two-arm randomized controlled clinical trial (RCT). The aims of this study are to compare the effectiveness of the BST (Brief Strategic Therapy) with the gold standard CBT (Cognitive Behavior Therapy) in a inpatient and telephone-based outpatient program in a sample of obese people with BED (Binge Eating Disorder) seeking treatment for weight reduction.

DETAILED DESCRIPTION:
Obesity constitutes one of the most important medical and public health problems of our time. It is considered as a chronic pathology and is widely recognized as a risk factor for many medical complications such as cardiovascular, orthopedic, pneumological and endocrinological diseases. Overweight and obesity is also linked with Binge Eating Disorder (BED). Binge eating disorder is characterized by frequent and persistent episodes of binge eating accompanied by feelings of loss of control and marked distress in the absence of regular compensatory behaviors. Functional interventions for significantly reduce weight, maintain weight loss and manage associated pathologies like BED are typically combined treatment options (dietetic, nutritional, physical, behavioral, cognitive-behavioral, pharmacological, surgical). Significant difficulties with regard to availability, costs, treatment adherence and long-term efficacy are present. Moreover most overweight and obese individuals regain about one third of the weight lost with treatment within 1 year [11] and they are typically back to baseline in 3 to 5 years.

Treatment for BED is directed towards either the physical or psychopathological impairments and Cognitive behavior therapy (CBT) and Interpersonal Psychotherapy (IPT) are psychotherapies for BED indicated to target the eating disorder. Particularly CBT is the therapeutic approach indicated both in inpatient and in outpatient settings for BED. In recent years systemic and systemic-strategic psychotherapies have been implemented to treat patients with obesity and BED involved in familiar problems. Particularly a brief protocol for the systemic-strategic treatment of BED, using overall the strategic dialogue, has been developed by Nardone and Portelli in the Handbook of Brief Strategic Therapy (BST).

Moreover telemedicine, a new promising low cost method, has been used for obesity with BED in outpatient settings in order to avoid relapses after the inpatient step of treatment and to keep on a continuity of care with to the involvement of the same clinical inpatient team.

For these reasons, we developed STRATOB (Systemic and STRATegic psychotherapy for OBesity), a comprehensive two-phase stepped down program enhanced by telepsychology for the medium-term treatment of obese people with BED seeking intervention for weight loss. The core aspects of STRATOB are the hospital-based intensive treatment and the continuity of care at home using a low-level of telecare (mobile phones). Many treatments delivered using technologies such as web-sites, e-mails, chat lines, videoconferences, UMTS-based mobile-phones and telephones) could be a valid integration to traditional psychotherapy reducing expensive and time-consuming clinical visits and improving adherence to prescribed psychological, dietetic and medical treatments through extensive monitoring and support.

This paper describes the design of the STRATOB study, a two-arm randomized controlled clinical trial (RCT). The aims of this study are to compare the effectiveness of the BST with the gold standard CBT in a inpatient and telephone-based outpatient program in a sample of obese people with BED seeking treatment for weight reduction.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years;
2. obesity according to the WHO criteria (BMI≥30)
3. BED (DSM-IV-TR criteria)
4. written and informed consent to participate

Exclusion Criteria:

1. other severe psychiatric disturbance diagnosed by DSM-IV-TR criteria
2. concurrent medical condition not related to obesity.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Psychological wellbeing | 6 months
  The Outcome Questionnaire (OQ 45.2) - Italian translation and validation The OQ 45.2 is an self report questionnaire developed by Michael Lambert in 1996. The OQ 45 items version is a measure of outcome and it is designed in order to collect repeated measures of patient progress during psychotherapy and after its conclusion. This instrument is one of the most used in psychotherapy research in the U.S. The OQ 45.2 is composed by 45 items that form 3 scales: Symptom Distress (SD), Interpersonal Relations (IR) e Social Role (SR), and a Global Index.

SECONDARY OUTCOMES:
Number of binge days in the week (assessed by self-report procedures) | 6 months
  The use of binge days in the week rather than binge episodes relates to the phenomenology of binge eating for patients with BED.

REFERENCES:
- [Derived] Jackson JB, Pietrabissa G, Rossi A, Manzoni GM, Castelnuovo G. Brief strategic therapy and cognitive behavioral therapy for women with binge eating disorder and comorbid obesity: A randomized clinical trial one-year follow-up. J Consult Clin Psychol. 2018 Aug;86(8):688-701. doi: 10.1037/ccp0000313. PMID 30035585
- [Derived] Castelnuovo G, Manzoni GM, Villa V, Cesa GL, Pietrabissa G, Molinari E. The STRATOB study: design of a randomized controlled clinical trial of Cognitive Behavioral Therapy and Brief Strategic Therapy with telecare in patients with obesity and binge-eating disorder referred to residential nutritional rehabilitation. Trials. 2011 May 9;12:114. doi: 10.1186/1745-6215-12-114. PMID 21554734